CLINICAL TRIAL: NCT01741129
Title: Comparison of Effectiveness of Nasal CPAP and Nasal IMV in Early Rescue Surfactant Treatment in Preterm Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mehmet Yekta (Other)
Responsible Party: Sponsor-Investigator, Mehmet Yekta, Zekai Tahir Burak Maternity and Teaching Hospital, Ankara, Zekai Tahir Burak Women's Health Research and Education Hospital
Organization: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZTB2611
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2013-01

CONDITIONS: Noninvasive Ventilation for Respiratory Distress Syndrome
Keywords: Nasal CPAP; Nasal IMV; Surfactant; Preterm infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal Continuous Positive Airway Pressure (CPAP) (Active Comparator): After 2 hours evaluation:
  * Infants needed invasive MV (mechanic ventilation) or Required a fraction of inspired oxygen of >40% to maintain the targeted saturation of >88% to 92%.
  * Non-invasive surfactant treatment (Curosurf®) 100 mg/kg per dose
  Interventions: Device: Nasal CPAP (SLE)
- Nasal Intermittent Mandatory Ventilation (IMV) (Active Comparator): After 2 hours evaluation:
  * Infants needed invasive MV or Required a fraction of inspired oxygen of >40% to maintain the targeted saturation of > 88% to 92%.
  * Non-invasive surfactant treatment (Curosurf®) 100 mg/kg per dose
  Interventions: Device: Nasal IMV (SLE)

INTERVENTIONS:
Device: Nasal CPAP (SLE) — PEEP: 4-6 cmH2O, Flow: 8 to 10 L/minute
  Other Names: SLE 2000, SLE 5000
  Arms: Nasal Continuous Positive Airway Pressure (CPAP)
Device: Nasal IMV (SLE) — PIP: 15-20 cmH2O, PEEP: 4-6 cmH2O, Inspiratory time: 0.4-0.5 second, Rate: 20-30 /minute
  Other Names: SLE 2000, SLE 5000
  Arms: Nasal Intermittent Mandatory Ventilation (IMV)

SUMMARY:
The investigators aimed to compare the efficacy of nasal intermittent mandatory ventilation (IMV) and nasal continuous positive airway pressure (CPAP) in early rescue surfactant treatment in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

- Gestational age 26-32 weeks

The criteria for failure were met by at least 1 of the following:

* pH: 7.10 and PaCO2: 70 mm Hg
* Recurrent apnea with >3 episodes (Prophylactic caffeine were used in all infants)
* Single episode of apnea that required bag-and-mask ventilation
* PaO2: 50 mmHg with a fraction of inspired oxygen of >0.5.

Exclusion Criteria:

* Major congenital anomalies
* Presence of cardiovascular instability
* Intubation at admission to the NICU
* Consent not provided or refused

Max Age: 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of nasal intermittent mandatory ventilation (IMV) and nasal continuous positive airway pressure (CPAP) in early rescue surfactant treatment in preterm infants | 3 months
  If infants needed invasive MV or Required a fraction of inspired oxygen of >40% to maintain the targeted saturation of >88% to 92%, surfactant treatment will give for respiratory distress syndrome (RDS). It means that nasal IMV or CPAP is ineffective.

SECONDARY OUTCOMES:
Complications of respiratory support | 3 months
  respiratory insufficiency, pneumothorax

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Oncel MY, Arayici S, Uras N, Alyamac-Dizdar E, Sari FN, Karahan S, Canpolat FE, Oguz SS, Dilmen U. Nasal continuous positive airway pressure versus nasal intermittent positive-pressure ventilation within the minimally invasive surfactant therapy approach in preterm infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2016 Jul;101(4):F323-8. doi: 10.1136/archdischild-2015-308204. Epub 2015 Nov 9. PMID 26553376